CLINICAL TRIAL: NCT06593704
Title: Proactive Population Health Management of Cardiovascular Disease in Primary Care Using a Multilevel Guideline Adherence Toolkit (the PROSPERA-program).
Brief Title: Proactive Population Health Management of Cardiovascular Disease in Primary Care Using the PROSPERA-program.
Acronym: PROSPERA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Principal Investigator, rcvos, Principal Investigator R.C. Vos, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-3050; 10140302110018 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases
Keywords: Primary Care; Population Health Management; Implementation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROSPERA (Experimental): The PROSPERA-program
  Interventions: Other: PROSPERA-program
- Control (No Intervention): Primary cardiovascular care-as-usual, according to national and international applicable guidelines.

INTERVENTIONS:
Other: PROSPERA-program — The PROSPERA-program consists of the following components:
  1. Health care provider training and education about U-Prevent and cardiovascular risk communication.
  2. Risk stratification: proactive selection of cardiovascular patients through the PROSPERA-empanelment procedure - for the population with increased cardiovascular risk, prior to consultation.
  3. Decision support tools: use of the Lifestylecheck and the U-Prevent clinical decision support tool to guide motivated shared decision making towards appropriate care matched to the care complexity of the patient - for the individual patient, during consultation.
  Arms: PROSPERA

SUMMARY:
The PROSPERA-program is a complex multilevel approach that includes training for healthcare providers, a risk assessment process, and decision support tools to help match patients with the appropriate treatment based on their care needs.

The goal of this clinical trial is to determine if the PROSPERA-program can improve the cardiovascular risk profile in patients aged 40-90 years enrolled in primary care programs for increased cardiovascular risk, such as cardiovascular disease, increased vascular risk, or diabetes.

The main question it aims to answer is:

• Does the cardiovascular risk profile improve for patients using the PROSPERA-program?

Researchers will compare the PROSPERA-program with standard cardiovascular care to see if the program enhances cardiovascular population health in primary care.

Additionally, the study will assess how well the PROSPERA-program fits into the workflow of primary care providers and supports shared decision-making.

Participants will:

* Receive a consultation with their general practitioner or practice nurse according to the PROSPERA-program.
* Have their routinely collected healthcare data used for evaluation.
* Be asked to complete a questionnaire or participate in an interview (for a subset of patients).

ELIGIBILITY:
Inclusion criteria:

* Age > 40 years and ≤ 90 years
* Patient in a primary care practice enrolled in this study
* Included in the cardiovascular disease (CVD), increased vascular risk (IVR) or diabetes mellitus (DM) Dutch Integrated Care programs
* Additional criteria for subgroup that receives questionnaires: able to communicate in the Dutch and/or English language

Exclusion Criteria:

* Patients with Diabetes Mellitus type I
* Patients receiving palliative care
* Patients with any form of cognitive impairment diseases such as Dementia or Alzheimer
* Patients who are treated in other Integrated Care programs because of their frailty (e.g. elderly who are treated in the 'Kwetsbare Ouderen Chronische Zorgprogramma')

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 848 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-07-09 (Estimated); Study Completion 2026-07-09 (Estimated)

PRIMARY OUTCOMES:
The proportion of individuals who have achieved all protocol-defined cardiovascular prevention goals. | At 0 and 18 months
  Protocol-defined treatment goals are in line with local prevention targets (including treatment targets such as Systolic Blood Pressure, LDL-cholesterol, Antithrombotic therapy, HbA1c, SGTL2 inhibitors and/or GLP1-receptor agonists).
  The sample size is based on the minimum number of subjects (patients) who will complete the component of the intervention conducted during consultation (= the clinical decision tools). A subset will receive additional questionnaires.
  The primary outcome will be compared among the complete study population as well as in the subgroup.

SECONDARY OUTCOMES:
Perceived shared decision making (in subset only) | immediately after the intervention
  9-item Shared Decision Making Questionnaire (SDM-Q-9)
Perceived shared decision making (in subset only) | immediately after the intervention
  Patient interviews (qualitative)
Decisional Conflict (in subset only) | immediately after the intervention
  The Decisional Conflict Scale (DCS)
Implementation outcome: fidelity | At month 4 and 10
  Percentage of target population that has received the U-Prevent component of the PROSPERA-program during the study duration as measured by the U-Prevent logbook.
Implementation outcome: fidelity | At month 4 and 10
  Fidelity checklist by HCPs
  .
Implementation outcome: penetration | At month 10
  The number of health care professionals who deliver the PROSPERA-program on an individual patient level (component 2) divided by the number of health care professionals who are expected to deliver this service.
Healthcare professional's satisfaction on usability of the PROSPERA-program | At month 10
  System Usability Scale
Cost-effectiveness | immediately after the intervention and at month 18
  Cost-effectiveness of the PROSPERA-program in Quality-Adjusted Life Years (QALYs) as calculated in a cost-effectiveness analysis

CONTACTS AND LOCATIONS:
Overall Officials: Rimke C Vos, Principal Investigator — LUMC; Mattijs E Numans, Principal Investigator — LUMC; Jannick AN Dorresteijn, Principal Investigator — UMC Utrecht; Hendrikus JA van Os, Principal Investigator — LUMC
Locations (1):
- Department of Public Health and Primary Care, The Hague, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Due to the nature of the study, blinding is not possible. Therefore, the data might contain privacy sensitive information and only restricted access can be granted for parts of the collected data. It has yet to be decided which data can be acquired through restricted access.